CLINICAL TRIAL: NCT03485092
Title: Studies of Empagliflozin and Its Cardiovascular, Renal and Metabolic Effects in Patients With Diabetes Mellitus (or Pre-diabetes) and Heart Failure (SUGAR-DM-HF)
Brief Title: Studies of Empagliflozin and Its Cardiovascular, Renal and Metabolic Effects
Acronym: SUGAR-DM-HF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GN15CA580
Record Dates: First submitted 2018-03-19; First posted 2018-04-02 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Heart Failure; Diabetes Mellitus
Keywords: heart failure; diabetes mellitus; empagliflozin; Randomised, placebo controlled trial
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Randomised, placebo controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: placebo controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin (Active Comparator): Empagliflozin 10mg tablets for oral self-administration once daily
  Interventions: Drug: Empagliflozin 10 MG
- Placebo Oral Tablet (Placebo Comparator): placebo tablets for oral self-administration once daily
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Empagliflozin 10mg tablets for oral self administration once a day
  Arms: Empagliflozin
Drug: Placebo Oral Tablet — placebo tablets for oral self administration once a day
  Arms: Placebo Oral Tablet

SUMMARY:
The investigators hypothesise that empagliflozin 10mg daily will have haemodynamic, cardiac, and renal benefits compared to placebo over 36 weeks in heart failure patients with type 2 diabetes (or pre-diabetes), leading to measurable improvements in clinical measures of cardiac structure and function (LVESVI, and LV strain) as well as renal blood flow.

DETAILED DESCRIPTION:
The results of the EMPA-REG OUTCOME trial on CVD outcomes and heart failure hospitalisation suggests that empagliflozin works quickly to lessen CVD mortality and reduce heart failure hospitalisations in patients with diabetes and existing cardiovascular disease. The lack of effect on non-fatal MI and stroke would suggest limited impact on atherothrombotic mechanisms. It is important to understand the mechanisms by which empagliflozin is acting in more detail, in order that the drug can be more widely targeted at patient groups that might benefit most; particularly patients with heart failure and diabetes (or pre-diabetes) (as discussed in the rationale).

The investigators have hypothesised, in a detailed published review, that the benefit derives from the specific effects of sodium-glucose linked transporter-2 (SGLT2) inhibition on renal sodium and glucose handling, leading to both diuresis and improvements in diabetes-related maladaptive renal arteriolar responses. These haemodynamic and renal effects are likely to be beneficial in patients with clinical or subclinical cardiac dysfunction. The net result of these processes is an improvement in cardiac systolic and diastolic function and, thereby, a lower risk of heart failure hospitalisation (HFH) and sudden cardiac death.

The investigators have therefore designed the present trial to perform a comprehensive clinical trial to interrogate in detail the effects of empagliflozin on specific pathways (inclusive of cardiac and renal effects) in patients with type 2 diabetes (or pre-diabetes) and heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male or female, aged ≥18 years age
* Type 2 DM (diet-controlled or on stable treatment) or prediabetes

  * Stable treatment defined as no change in oral therapy agents or doses for diabetes mellitus and (where applicable) <10% change in average total daily insulin dose over last 6 weeks
  * HbA1c ≤97 mmol/mol (11%) (routine available data from medical records, recorded in the last year)
  * Prediabetes defined as HbA1c 39-47 mmol/mol (5.7-6.4%) at the time of screening (specifically for the prediabetes group, HbA1c will be repeated at the time of screening if there are no recent results within the last 3 months, in order to confirm the diagnosis of prediabetes)
* Heart failure (as defined by the presence of typical signs and symptoms of heart failure with documented reduced ejection fraction (ref SIGN and ESC guidelines))

  * NYHA class II-IV
  * LVEF ≤40%
  * On stable doses of ACEI, ARB or ARNI for 4 weeks prior to randomisation unless contraindicated or not tolerated. They should also be taking a beta-blocker at a stable dose for 4 weeks unless contraindicated or not tolerated
* Women of childbearing potential (WOCBP) must be currently adhering to, or be willing to use, highly effective birth control methods for study treatment duration including:

  * Combined hormonal contraception (oestrogen and progestogen containing medication) either orally, intravaginally, or transdermally
  * Progesterone only hormonal contraception either orally, injected, or implanted
  * Intrauterine device (IUD)
  * Intrauterine hormone release system (IUS)
  * Bilateral fallopian tube occlusion
  * Vasectomised partner
  * Complete sexual abstinence where this is their preferred and usual lifestyle

WOCBP comprises women who have experienced menarche and who have not undergone successful surgical sterilisation (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or who are not post-menopausal. Post-menopausal is defined as:

o Women who have had amenorrhea for ≥12 consecutive months (without another medical cause)

Exclusion Criteria:

* Type 1 DM
* History of hospital admission with a diagnosis of diabetic ketoacidosis (DKA)
* Insulin use within 1 year of diagnosis of diabetes
* History of acute or chronic pancreatitis
* eGFR <30 ml/min/1.73m2 (derived using CKD EPI)
* Persistent/permanent atrial fibrillation/flutter (conditions which significantly impede MRI image interpretability)
* Acute coronary syndrome, stroke or surgery within 1 month (small type 2 MI in the context of acute HF does not apply)
* BMI >52 kg/m2
* Liver disease, defined by serum levels of alanine aminotransferase, aspartate aminotransferase, or alkaline phosphatase above 3 x upper limit of normal (ULN) during screening
* Bariatric surgery within the past two years and other gastrointestinal surgeries that induce chronic malabsorption
* Any condition outside the cardiovascular and renal disease area, such as but not limited to malignancy, with a life expectancy of less than 2 years based on investigator's clinical judgement
* Active malignancy requiring treatment at the time of visit 1 (with the exception of successfully treated basal cell or treated squamous cell carcinoma, adjuvant hormonal therapy for breast cancer and hormone therapy for prostate cancer)
* Blood dyscrasias or any disorders causing haemolysis or unstable red blood cells (e.g. malaria, babesiosis, haemolytic anaemia)
* Treatment with systemic steroids at time of informed consent or change in dosage of thyroid hormones within 6 weeks prior to informed consent
* Any uncontrolled endocrine disorder except Type 2 DM
* Alcohol or drug abuse within 3 months of informed consent that would interfere with trial participation or any ongoing condition leading to decreased compliance with study procedures or study drug intake
* Known hypersensitivity to the empagliflozin or excipients
* Known hypersensitivity to gadolinium
* Inability to give informed consent
* SGLT2 inhibitor use (current or previous)
* Devices or any other contraindication to MRI scans
* Currently pregnant, planning pregnancy, or currently breastfeeding
* History of previous lower limb amputation
* Current participation in another interventional medical study or within the last 90 days
* Anyone who, in the investigators' opinion, is not suitable to participate in the trial for other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2020-03-28 (Actual); Study Completion 2020-03-28 (Actual)

PRIMARY OUTCOMES:
Left Ventricular End Systolic Volume Index (LVESVI) | 36 weeks
  Cardiac structure measured by left ventricular end-systolic volume index measured by cardiac magnetic resonance imaging as mL/m2
left ventricular global longitudinal strain (GLS) | 36 weeks
  Cardiac structure measured by left ventricular global longitudinal strain measured by cardiac magnetic resonance imaging GLS%

SECONDARY OUTCOMES:
Left ventricular end diastolic volume index (LVEDVI) | 36 weeks
  Left ventricular end diastolic volume index (LVEDVI) measured by Cardiac MR in ml/m2
Left ventricular ejection fraction (LVEF) | 36 weeks
  Left ventricular ejection fraction (LVEF) measured by Cardiac MR in percentage
Left ventricular mass index (LVMI) | 36 weeks
  Left ventricular mass index (LVMI) measured by cardiac MR in grams/m2
Left ventricular global function index (LVGFI) | 36 weeks
  Left ventricular global function index (LVGFI) measured by cardiac MR in percentage
Left atrial volume index (LAVI) | 36 weeks
  Left atrial volume index (LAVI) measured by cardiac MR in ml/m2
Microvascular perfusion | 36 weeks
  Microvascular perfusion measured by Gadolinium enhanced Cardiac magnetic resonance imaging measured as ml/min/g
Extracellular volume fraction | 36 weeks
  Extracellular volume fraction measured by Gadolinium enhanced Cardiac magnetic resonance imaging measured as %
Kansas City Cardiomyopathy Questionnaire (KCCQ) Total Symptom Score (TSS) | 36 weeks
  Kansas City Cardiomyopathy Questionnaire Total Symptom score (TSS) measured by mean overall difference and responder analysis (higher score = better outcome)
6 minute walk distance (Exercise Capacity) | 36 weeks
  Exercise capacity measured by six minute walk test measured in m
Pulmonary congestion | 36 weeks
  Pulmonary congestion as B-lines measured using lung ultrasound
Biomarker profile -glycated haemaglobin (HbA1c) | 36 weeks
  biomarker profile of HbA1c (mmol/mol)
Biomarker profile - creatine | 36 weeks
  biomarker profile of creatine (umol/L)
Biomarker profile - estimated glomerular filtration rate (eGFR) | 36 weeks
  biomarker profile of eGFR (ml/min/m2)
Biomarker profile - liver function tests (LFTs) | 36 weeks
  biomarker profile of LFTs (U/L)
Biomarker profile - uric acid | 36 weeks
  biomarker profile of uric acid (umol/L)
Intensification of diuretic therapy | 36 weeks
  Intensification of diuretic therapy through addition and/or increase dose of diuretic medication

OTHER OUTCOMES:
Left ventricular global longitudinal strain (GLS) | 36 weeks
  Left ventricular global longitudinal strain (GLS) measured by CMR tagging measured in percentage
Left ventricular global circumferential strain (GCS) | 36 weeks
  Left ventricular global circumferential strain (GCS) measured in CMR featured-tracking and tagging in percentage
Left ventricular global radial strain (GRS) | 36 weeks
  Left ventricular global radial strain (GRS)measured in CMR featured-tracking and tagging in percentage
total renal blood flow measured by magnetic resonance imaging | 36 weeks
  total renal blood flow measure using cardiac magnetic resonance imaging measured as ml/min/100g
Renal fibrosis | 36 weeks
  Renal fibrosis measured by T1 mapping in MRI in miiliseconds
Bioelectrical impedance analysis | 36 weeks
  Bioelectrical impedance analysis in percentage
Clinical composite outcome of death, hospitalisation with worsening heart failure, ED visit for worsening heart failure, outpatient worsening of heart failure accompanied by increase in HF therapy | 36 weeks
  Clinical composite outcome of death, hospitalisation with worsening heart failure, ED visit for worsening heart failure, outpatient worsening of heart failure accompanied by increase in HF therapy
Clinical composite analysed using Win-ratio approach | 36 weeks
  Clinical composite (analysed using Win-ratio approach) outcome of death, hospitalisation with worsening heart failure, ED visit for worsening heart failure, outpatient worsening of heart failure accompanied by increase in HF therapy, KCCQ-TSS >5-point decrease, or no decrease, >30% in NT-proBNP from baseline
Left ventricular diastolic function | 36 weeks
  Left ventricular diastolic function measured by echocardiogram
DNA and epigenetics | 36 weeks
  DNA and epigenetic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Naveed Sattar, PhD, Study Chair — Glasgow University and NHS GGC
Locations (1):
- Queen Elizabeth University Hospital, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zinman B, Wanner C, Lachin JM, Fitchett D, Bluhmki E, Hantel S, Mattheus M, Devins T, Johansen OE, Woerle HJ, Broedl UC, Inzucchi SE; EMPA-REG OUTCOME Investigators. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2117-28. doi: 10.1056/NEJMoa1504720. Epub 2015 Sep 17. PMID 26378978
- [Derived] Kanie T, Mizuno A, Takaoka Y, Suzuki T, Yoneoka D, Nishikawa Y, Tam WWS, Morze J, Rynkiewicz A, Xin Y, Wu O, Providencia R, Kwong JS. Dipeptidyl peptidase-4 inhibitors, glucagon-like peptide 1 receptor agonists and sodium-glucose co-transporter-2 inhibitors for people with cardiovascular disease: a network meta-analysis. Cochrane Database Syst Rev. 2021 Oct 25;10(10):CD013650. doi: 10.1002/14651858.CD013650.pub2. PMID 34693515
- [Derived] Lee MMY, Brooksbank KJM, Wetherall K, Mangion K, Roditi G, Campbell RT, Berry C, Chong V, Coyle L, Docherty KF, Dreisbach JG, Labinjoh C, Lang NN, Lennie V, McConnachie A, Murphy CL, Petrie CJ, Petrie JR, Speirits IA, Sourbron S, Welsh P, Woodward R, Radjenovic A, Mark PB, McMurray JJV, Jhund PS, Petrie MC, Sattar N. Effect of Empagliflozin on Left Ventricular Volumes in Patients With Type 2 Diabetes, or Prediabetes, and Heart Failure With Reduced Ejection Fraction (SUGAR-DM-HF). Circulation. 2021 Feb 9;143(6):516-525. doi: 10.1161/CIRCULATIONAHA.120.052186. Epub 2020 Nov 13. PMID 33186500